CLINICAL TRIAL: NCT05158413
Title: High and Low Dose Oral Sesame Immunotherapy - Comparison of Efficacy and Safety
Acronym: Sesame
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sesame Protocol
Record Dates: First submitted 2021-11-24; First posted 2021-12-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
Keywords: sesame; food allergy; immunotherapy; children
MeSH Terms: conditions — Food Hypersensitivity; SeSAME syndrome | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups. During the maintenance phase, the first group will receive low dose of sesame protein, which amounts 300mg, the second will get high dose, which is 1200 mg of sesame protein. Oral immunotherapy with low (300mg) and high (1200mg) dose of sesame protein in children randomly assigned to two groups (1:1). Patients will receive ground sesame mixed with apple mousse (supposing apple tolerance). For the transparency of the study all patients will receive the same commercially prepared apple muss product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Experimental): Experimental: high dose of sesame 20 patients
  Interventions: Dietary Supplement: High dose
- Low dose (Active Comparator): Active Comparator: low dose of sesame 20 patients
  Interventions: Dietary Supplement: Low dose

INTERVENTIONS:
Dietary Supplement: High dose — Patients will receive a high dose of sesame paste or flour (1200 mg of sesame protein) mixed with apple mousse (supposing child tolerates apple). For the transparency of the study all patients will receive the same commercially prepared apple product
  Arms: High dose
Dietary Supplement: Low dose — Patients will receive a low dose of sesame paste or flour (300 mg of sesame protein) mixed with apple mousse (supposing child tolerates apple). For the transparency of the study all patients will receive the same commercially prepared apple product
  Arms: Low dose

SUMMARY:
In this trial the investigators aim to assess the effectiveness and safety of oral immunotherapy with sesame protein in high and low dose (300mg versus 1200mg) in children with sesame allergy.

DETAILED DESCRIPTION:
Sesame allergy is an important global clinical problem affecting 0,2-0,8% population. In food allergy, allergen avoidance and emergency treatment are still therapeutic hallmarks. Oral and sublingual allergen-specific immunotherapies have been provided as a new approach to managing food allergy. The main goal of oral immunotherapy is to obtain the desensitization to food. The oral immunotherapy (OIT) is considered as safe and highly effective, according to current research. In addition, this type of therapy reduce the influence of food allergy in patient's live.

Children 4 to 17 years old with sesame allergy will be enrolled into study. Skin prick test with condiment made from toasted ground hulled sesame and open oral food challenge (OOFC) will be performed at the baseline and at the end of procedure. Blood will be analyzed for specific IgE, IgG4 levels and basophil activation test before and after OIT. OIT will consisted of two parts: dosage increase phase and maintenance phase. The Participants will be randomized (1:1) to receive sesame OIT with maintenance dose of 300 mg or 1200 mg sesame protein.

In the dosage increase phase, the dose of condiment made from toasted ground hulled sesame will be gradually increased every two weeks and administrated to a child during hospitalization (1-day procedure). Precondition to increase of dose is good tolerance of previous portion of condiment made from toasted ground hulled sesame. The maximum time frame for this phase is 14 months.

After achieving tolerance, immunotherapy will be continued for 3 months in maintenance phase, with dose 300mg or 1200 mg sesame protein. Maintenance dose is determined by random patients' assignment to one from study's .

After 3 months (12 weeks +/-2 weeks) of maintenance dose the final OOFC and evaluation of desensitization of sesame protein will be performed. Confirmation of the total desensitization to sesame is the tolerance of a single dose of 4000 mg sesame protein.

ELIGIBILITY:
Inclusion Criteria:

* medical history of sesame allergy,
* IgE-mediated sesame allergy confirmed as positive skin prick tests with sesame allergens (diameter of the wheal greater than 3mm) and/or specific IgE level greater than 0.35 kilo units of Allergen per liter (kUA/l) (UniCAP method),
* reaction to sesame protein during OOFC (maximum dose 4000g),
* signed Informed Consent by parent/legal guardian and patient aged >16 years old,
* patient's/caregivers' cooperation with researcher.

Exclusion Criteria:

* no confirmed sesame allergy,
* negative oral food challenge with sesame protein (maximum dose 4000g),
* severe asthma,
* uncontrolled mild/moderate asthma: forced expiratory volume at one second (FEV1)<80% (under 5. percentile), FEV1/forced vital capacity (FVC)<75% (under 5. percentile), hospitalization due to asthma exacerbation within last 12 months,
* current oral/sublingual/subcutaneous immunotherapy with other allergen,
* eosinophilic gastroenteritis,
* a history of severe recurrent anaphylaxis episodes,
* chronic diseases requiring continuous treatment, including heart disease, epilepsy, metabolic diseases, diabetes,
* medication:

  * oral, daily steroid therapy longer than 1 month within last 12 months,
  * at least two courses of oral steroid therapy (at least 7 days) within last 12 months,
  * oral steroid therapy longer than 7 days within last 3 months,
  * biological treatment,
  * the need to constantly take antihistamines,
  * therapy with β-blockers, angiotensin converting enzyme (ACE) inhibitors, calcium channel inhibitors,
  * pregnancy,
  * no consent to participate in the study,
  * lack of patient cooperation.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tolerance of sesame | Up to 16 months after starting oral immunotherapy
  Proportion of participants who tolerate the single dose of 4000mg sesame protein

SECONDARY OUTCOMES:
Adverse event | Up to 16 months after starting oral immunotherapy
  Quantity and severity of adverse effect, assessed and compared between groups, divided into mild, moderate and severe category
Laboratory data | Up to 16 months after starting oral immunotherapy
  Difference in sesame serum immunoglobulin E (IgE) level and immunoglobulin G4 (IgG4) level, compared between groups at the end of treatment
Basophil activation test | Up to 16 months after starting oral immunotherapy
  The basophil activation test (BAT) results compared between groups at the end of treatment
Skin prick test (SPT) | Up to 16 months after starting oral immunotherapy
  Change in skin prick test reactivity to sesame protein from baseline to end of treatment, compared between groups
Desensitization dose | Up to 16 months after starting oral immunotherapy
  Change in maximum tolerated dose of sesame in oral food challenge before and in the end of treatment, compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grzela, MD, PhD, Study Chair — Medical University of Warsaw
Locations (1):
- Katarzyna Grzela, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta RS, Warren CM, Smith BM, et al. The Public Health Impact of Parent-Reported Childhood Food Allergies in the United States. Pediatrics. 2018:142(6):e20181235. Pediatrics. 2019 Mar;143(3):e20183835. doi: 10.1542/peds.2018-3835. No abstract available. PMID 30819972
- [Background] Gupta RS, Warren CM, Smith BM, Jiang J, Blumenstock JA, Davis MM, Schleimer RP, Nadeau KC. Prevalence and Severity of Food Allergies Among US Adults. JAMA Netw Open. 2019 Jan 4;2(1):e185630. doi: 10.1001/jamanetworkopen.2018.5630. PMID 30646188
- [Background] Dalal I, Goldberg M, Katz Y. Sesame seed food allergy. Curr Allergy Asthma Rep. 2012 Aug;12(4):339-45. doi: 10.1007/s11882-012-0267-2. PMID 22610362
- [Background] Warren CM, Chadha AS, Sicherer SH, Jiang J, Gupta RS. Prevalence and Severity of Sesame Allergy in the United States. JAMA Netw Open. 2019 Aug 2;2(8):e199144. doi: 10.1001/jamanetworkopen.2019.9144. PMID 31373655
- [Background] Nachshon L, Goldberg MR, Levy MB, Appel MY, Epstein-Rigbi N, Lidholm J, Holmqvist M, Katz Y, Elizur A. Efficacy and Safety of Sesame Oral Immunotherapy-A Real-World, Single-Center Study. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2775-2781.e2. doi: 10.1016/j.jaip.2019.05.031. Epub 2019 May 29. PMID 31150789
- [Background] Adatia A, Clarke AE, Yanishevsky Y, Ben-Shoshan M. Sesame allergy: current perspectives. J Asthma Allergy. 2017 Apr 27;10:141-151. doi: 10.2147/JAA.S113612. eCollection 2017. PMID 28490893
- [Background] Brough HA, Caubet JC, Mazon A, Haddad D, Bergmann MM, Wassenberg J, Panetta V, Gourgey R, Radulovic S, Nieto M, Santos AF, Nieto A, Lack G, Eigenmann PA. Defining challenge-proven coexistent nut and sesame seed allergy: A prospective multicenter European study. J Allergy Clin Immunol. 2020 Apr;145(4):1231-1239. doi: 10.1016/j.jaci.2019.09.036. Epub 2019 Dec 20. PMID 31866098
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Feuille E, Nowak-Wegrzyn A. Allergen-Specific Immunotherapies for Food Allergy. Allergy Asthma Immunol Res. 2018 May;10(3):189-206. doi: 10.4168/aair.2018.10.3.189. PMID 29676066